CLINICAL TRIAL: NCT03423485
Title: A Prospective, Multi-center, Single-arm, Open-label Study Designed to Evaluate Safety and Performance Profile of the CG-100 Intraluminal Bypass Device in Patients Undergoing Colorectal Surgery
Brief Title: Safety and Performance of the CG-100 in Patients Undergoing Colorectal Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colospan Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLD-017
Record Dates: First submitted 2017-12-21; First posted 2018-02-06 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Surgery
Keywords: Colorectal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Anastomosis is performed according to Standard of Care with the addition of the CG-100 Intraluminal Bypass Device
  Interventions: Device: CG-100 Intraluminal Bypass Device

INTERVENTIONS:
Device: CG-100 Intraluminal Bypass Device — Intended to reduce contact of fecal content with an anastomotic site , following colorectal surgery.

SUMMARY:
The purpose of this study is to evaluate the CG-100 device, a single use, temporary intraluminal bypass device,intended to reduce contact of fecal content with an anastomotic site, following colorectal surgery (open or laparoscopic)

DETAILED DESCRIPTION:
Colospan is initiating a pivotal clinical prospective, multi-center, single-arm, open-label study designed to evaluate safety and performance profile of the CG-100 Intraluminal Bypass Device in patients undergoing colorectal surgery study.

Up to 137 patients (in total) will be enrolled in up to 12 sites in Europe, Israel and USA.

Study objectives Primary Objective: To evaluate the performance of the CG-100 Intraluminal Bypass Device, in reducing contact of fecal content with an anastomotic site in patients undergoing colorectal surgery (open, robotic, or laparoscopic) Secondary Objectives: To evaluate Performance in terms of clinical and radiological anastomotic leakage Successful positioning and maintenance of device position To assess the ease of the device's application and removal Safety: To assess the safety profile of the CG-100 Intraluminal Bypass Device.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is willing to comply with protocol-specified follow-up evaluations
2. Patient 22-75 years of age at screening
3. The patient is scheduled to undergo an elective colorectal surgery (open, laparoscopic, or robotic) which will require the creation of an anastomosis, maximally 20 cm proximal from the anal verge
4. The patient or legally authorized representative, has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the appropriate Medical Ethics Committee (EC) or Institutional Review Board (IRB).

Exclusion Criteria:

Preoperative

1. Pregnant or nursing female subjects. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to surgical procedure per site standard test.
2. Patient surgical treatment is acute (not elective)
3. Patient has local or systemic infection at the time of intervention (e.g., peritonitis)
4. Major surgical or interventional procedures within 30 days prior to this study or planned surgical or interventional procedures within 30 days of entry into this study
5. Patients with ASA classification > 3
6. Albumin < 30 g/liter
7. Patient has a diagnosis of bowel obstruction, bowel strangulation, peritonitis, bowel perforation, ischemic bowel, carcinomatosis or extensively spread inflammatory bowel disease
8. BMI ≥ 40
9. Subject is going through another surgical procedure (other than ileostomy or adhesiolysis) during the surgery.
10. Patient is participating in another clinical trial within 30 days of screening
11. Patient has been taking regular steroid medication in the last 6 months.
12. Patient has contraindications to general anesthesia
13. Patient has preexisting sphincter problems
14. Patient has evidence of extensive local disease in the pelvis
15. Any condition which in the opinion of the investigator may jeopardize the patient's safe participation Intraoperative (prior to device deployment)
16. Anastomosis is located more than 20 cm from the anal verge
17. Internal diameter lumen of the colon is smaller than 25 mm or larger than 34 mm
18. Blood loss (> 500 cc)
19. Anastomosis was not performed for any reason other than consequences as a result of use of the study device -

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the performance of the CG-100 Intraluminal Bypass Device, in reducing contact of fecal content with an anastomotic site in patients undergoing colorectal surgery (open, robotic, or laparoscopic) | device removal day (10 days +/-1)
  Leak proof seal with at least 85% success at balloon-Mucosa interface as evidenced by contrast through the device lumen without extravasation and no illumination of the anastomosis.

SECONDARY OUTCOMES:
To assess the safety profile of the CG-100 Intraluminal Bypass Device. | During surgical procedure and up to 30 days (+/- 5) ]
  Rate of adverse events
To evaluate Performance in terms of clinical anastomotic leakage based on clinical symptoms of the patient such as fever, blood tests. | Device deployment until device removal day (10 days +/-1)
  The patient will be followed for 10±1 days to assess the occurrence of clinical anastomotic leakage based on positive clinical symptoms of the patient such as fever, blood tests, while the CG-100 Intraluminal Bypass Device is in situ.
  In addition, at 10±1 days a rectal contrast enema will be done to assess the occurrence of radiological anastomotic leakage.
Successful positioning and maintenance of device position | 10+1 days post-surgery before device removal
  Position of internal sheath during rectal contrast enema based on radiological demonstration
To assess the ease of the device's application and removal | Surgical procedure and Device removal day (10 days +/-1)
  Assessment of the ease of the device's application will be done using a Device application use questionnaire completed by the surgeon at Procedure Day. The ease of device removal will also be assessed on Discharge Day, using the Device application use questionnaire
To assess the safety profile of the CG-100 Intraluminal Bypass Device. | Up to 30 (+/- 5) days
  Rate of device related complications
To assess the occurrence of radiological anastomotic leakage, evaluated by performing a rectal contrast enema . | At 10±1 days
  At 10±1 days a rectal contrast enema will be done to assess the occurrence of radiological anastomotic leakage.

CONTACTS AND LOCATIONS:
Overall Officials: Ilia Pinsk, MD, Principal Investigator — Soroka University Medical Center
Locations (5):
- Hospital Beaujon, Paris, Clichy, France
- University Hospital of Hamburg, Hamburg, Germany
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Carmel Medical Center, Haifa
- CHUV, University Hospital Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No